CLINICAL TRIAL: NCT00779454
Title: Combined Biological Treatment and Chemotherapy for Patients With Inoperable Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GOX-P; S-20080081; 2612-3769
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2016-06

CONDITIONS: Cholangiocarcinoma
Keywords: KRAS wild-type; Cholangiocarcinoma; Inoperable
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Oxaliplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KRAS wildtype (Other)
  Interventions: Drug: Panitumumab, Gemcitabine, Oxaliplatin, Capecitabine
- KRAS mutation (Other): Inclusion has been completed in the KRAS mutation arm.
  Interventions: Drug: Gemcitabine, Oxaliplatin, Capecitabine,

INTERVENTIONS:
Drug: Gemcitabine, Oxaliplatin, Capecitabine, — Gemcitabin: 1,000 mg/m2 day 1 Oxaliplatin: 60 mg/m2 day 1 Capecitabine: 1,000 mg/m2 x 2 daily days 1-7
  Arms: KRAS mutation
Drug: Panitumumab, Gemcitabine, Oxaliplatin, Capecitabine — Gemcitabine: 1,000 mg/m2 day 1 Oxaliplatin: 60 mg/m2 day 1 Capecitabine: 1,000 mg/m2 x 2 daily days 1-7 Panitumumab: 6 mg/kg day 1
  Arms: KRAS wildtype

SUMMARY:
The purpose of this study is partly to continue the good experience the investigators have with chemotherapy and partly to optimize treatment of inoperable cholangiocarcinoma by adding a biological antibody to the treatment of patients with wild-type Kirsten rat sarcoma viral oncogene homolog (KRAS).

DETAILED DESCRIPTION:
Cholangiocarcinoma is a relatively rare disease. In Denmark approximately 150 patients are diagnosed each year. A small part of the patients can be offered surgery, but the operation will rarely be radical, and most patients with cholangiocarcinoma are therefore candidates for chemotherapy.

In Denmark the combination therapy of Gemcitabine, Oxaliplatin and Capecitabine has been used in recent years. Based on experience with gastrointestinal tumors, however, there seems to be an effect of new biological substances, including EGFR antibodies. There are casuistic reports on the specific effect of a monoclonal antibody against EGFR in cholangiocarcinoma.

The effect of EGF is mediated through an intracellular pathway involving the KRAS protein. It has been shown that a mutation of KRAS causes the EGF system to be constantly activated. Effect in patients with a KRAS mutation is therefore not to be expected. Approximately 50% of the patients present this mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma arisen from gallbladder, extra or intrahepatic bile ducts or malignant cells consistent with the above and concomitant radiologic findings consistent with cholangiocarcinoma.
* Curative treatment presently discounted (surgery, stereotactic radiotherapy, etc.)
* KRAS analyzed and found wild-type (wt) or mutated
* PS 0-2
* Evaluable disease according to RECIST criteria, i.e., the disease does not need to be measurable
* Haematology:

  * ANC ≥ 1.5 x 10^9/l
  * Thrombocytes ≥ 100x10^9/l
* Biochemistry:

  * Bilirubinaemia ≤ 3 x upper normal value
  * ALAT ≤ 5 x upper normal value
* Creatinin ≤ upper normal value. If raised creatinin, the measured or calculated GFR must be at least 50% of the lower normal value.
* Fertile women must present a negative pregnancy test and use birth control during and 3 months after treatment. The following methods are considered safe birth control: Birth control pills, coil, gestagen deposit injection, subdermal implantation, hormonal vagina ring, and transdermal deposit band-aid)
* Oral and written informed consent

Exclusion Criteria:

* Chemotherapy within 4 weeks
* Radiotherapy within 4 weeks
* Immunotherapy within 4 weeks
* Other concomitant experimental treatment
* Known neuropathy ≥ grade 2
* Serious congruous medical disease
* Other previous malignant disease within 5 years, excl. non-melanoma skin cancer and carcinoma in situ cervicis uteri
* Previous serious and unexpected reactions to fluoropyrimidine treatment
* Hypersensitivity to one or more of the active substances, auxiliary substances or fluoruracil
* Patients with interstitial pneumonitis or pulmonary fibrosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to 6 months

SECONDARY OUTCOMES:
Response rate | 6 months
Overall survival | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Vejle Hospital, Vejle, Denmark
Locations (1):
- Vejle Hospital, Dept. of Oncology, Vejle, Denmark

REFERENCES:
- [Derived] Jensen LH, Andersen RF, Byriel L, Fernebro E, Jakobsen A, Lindebjerg J, Nottelmann L, Ploen J, Hansen TF. Phase II study of gemcitabine, oxaliplatin and capecitabine in patients with KRAS exon 2 mutated biliary tract cancers. Acta Oncol. 2020 Mar;59(3):298-301. doi: 10.1080/0284186X.2019.1701201. Epub 2019 Dec 14. PMID 31838939
- [Derived] Jensen LH, Lindebjerg J, Ploen J, Hansen TF, Jakobsen A. Phase II marker-driven trial of panitumumab and chemotherapy in KRAS wild-type biliary tract cancer. Ann Oncol. 2012 Sep;23(9):2341-2346. doi: 10.1093/annonc/mds008. Epub 2012 Feb 23. PMID 22367707